CLINICAL TRIAL: NCT02587013
Title: Randomized Controlled Trial of Uterine Exteriorization Versus in Situ Repair for Elective Cesarean Delivery
Brief Title: Comparison of Uterine Repair Methods for Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Valerie Zaphiratos, Clinical associate professor, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 151019
Record Dates: First submitted 2015-10-21; First posted 2015-10-27 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Complications; Cesarean Section

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- In situ uterine repair (Experimental): The uterus is repaired in situ within the abdominal cavity, without exteriorization; intra-abdominal repair
  Interventions: Procedure: Type A of uterine repair: In situ
- Exteriorization of the uterus (Active Comparator): The uterine incision is repaired with the exteriorization of the uterus; extra-abdominal repair
  Interventions: Procedure: Type B of uterine repair: Exteriorization

INTERVENTIONS:
Procedure: Type A of uterine repair: In situ — The uterine incision is closed with the uterus within the abdominal cavity
  Other Names: Intra-abdominal uterine repair
  Arms: In situ uterine repair
Procedure: Type B of uterine repair: Exteriorization — The uterine incision is repaired with the exteriorization of the uterus
  Other Names: Extra-abdominal uterine repair; Exteriorisation of the uterus
  Arms: Exteriorization of the uterus

SUMMARY:
This study is designed to compare the exteriorization of the uterus versus the in situ repair for closure of the hysterotomy incision with a completely standardized anesthetic protocol.

DETAILED DESCRIPTION:
Two well-known uterine repair techniques are described; the uterus can be repaired in situ within the peritoneal cavity (intraabdominal) or exteriorized temporarily from the abdomen for the closure of the hysterotomy incision (extraabdominal). 3 meta-analysis on the topic were unable to demonstrate the superiority of one technique regarding maternal morbidities. However, there is a paucity of studies with a standardized anesthetic protocol evaluating these outcomes.

This study will evaluate the impact of the uterine repair technique on different maternal morbidities; focusing on intra-operative nausea and vomiting under a standardized anesthetic protocol.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean delivery
* Term gestation, 37 weeks or more
* Healthy parturients (ASA 1 and 2)
* Spinal anesthesia

Exclusion Criteria:

* Conditions at risk of uterine atony and/or postpartum hemorrhage (multiple gestation, placenta accrete / previa, pre-eclampsia / eclampsia, uterine leiomyomata, polyhydramnios)
* Morbid obesity (BMI > 35 kg / m2) at delivery
* Coagulopathy
* Active labor
* Cardiomyopathy
* Emergency cesarean section
* Refusal/Inability to consent
* Language other than English or French

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Incidence of intraoperative nausea and vomiting | Intraoperative
  Incidence of intraoperative nausea and vomiting using a scale of 0 to 3; 0 being no nausea, 1 being light nausea, 2 being severe nausea, and 3 being nausea accompanied with vomiting and / or retching.
  The patients will be questioned at 5 pre-determined time points during the cesarean delivery.

SECONDARY OUTCOMES:
Incidence of hypotension | Intraoperative
  Hypotensive episodes, defined as a difference of more than 20% of the baseline mean arterial pressure, despite a phenylephrine infusion
Pelvic irrigation | Intraoperative
  To determine if the patient had pelvic irrigation, yes or no
Length of surgery | Intraoperative
Estimated blood loss | Intraoperative
  Measuring suction canisters and wet sponges
Reduction in hemoglobin | Within 24 hours of surgery
  Difference between preoperative and postoperative hemoglobin within 24 hours of surgery
Incidence of endometritis | Through study completion; on average of 1 year
Time to return of bowel function | Up to 2 weeks
  The return of bowel function will be assessed by listening to each of the four abdominal quadrants for intestinal peristalsis with a stethoscope twice a day and by assessing the time of the first gas or bowel movement. The first occurrence of any of these events will determine the return of intestinal transit.
Length of hospital stay after the cesarean delivery | Through study completion on average of 1 year
Incidence of tachycardia | Intraoperative
  Tachycardia, defined as a heart rate above 100 beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Zaphiratos, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Mireault D, Loubert C, Drolet P, Tordjman L, Godin N, Richebe P, Zaphiratos V. Uterine Exteriorization Compared With In Situ Repair of Hysterotomy After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2020 May;135(5):1145-1151. doi: 10.1097/AOG.0000000000003821. PMID 32282591